CLINICAL TRIAL: NCT06383325
Title: Evaluation of Liver Function Test to Identify Hepatotoxcicity Among Acute Leukemia Patients Who Are Receiving Chemotherapy Induction
Brief Title: Livertoxcicity in Acute Leukemia Patients During Chemotherapy Treatment
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Nada Hohamed Hamada Wahba, Doctor, Assiut University
Other Study IDs: Livertoxcicity in AL
Record Dates: First submitted 2024-04-22; First posted 2024-04-25 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Liver Toxicity, Chemically-Induced
MeSH Terms: conditions — Chemical and Drug Induced Liver Injury | interventions — Drug Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Combination Product: Chemotherapy — Detection of hepatotoxicity in acute leukemia patients during chemotherapy

SUMMARY:
Detection of hepatotoxcicity in acute leukemia and study the outcome of acute leukemia patients that suffer from hepatic toxiciyt

DETAILED DESCRIPTION:
Chemotherapy induction associated with hepatotoxicity during the induction has never been studied the study aimed to determine whether chemotherapy induction is associated with livertoxicity or not

ELIGIBILITY:
Inclusion Criteria:

* patients newly diagnosed with acute leukemia who are going to start chemotherapy treatment

Exclusion Criteria:

* patients previously diagnosed Acute leukemia and started treatment or in post treatment follow up

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Participants who will be diagnosed as acute leukemia and going to receive chemotherapy after
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Detection of hepatotoxcicity in acute leukemia during chemotherapy treatment | 3 months
  Evaluation of liver function test to identfy hepatotoxicity during chemotherapy treatment

REFERENCES:
- [Background] Mekonnen AT, Wondmeneh TG. Evaluation of liver function tests to identify hepatotoxicity among acute lymphoblastic leukemia patients who are receiving chemotherapy induction. Sci Rep. 2022 Aug 2;12(1):13215. doi: 10.1038/s41598-022-17618-w. PMID 35918381